CLINICAL TRIAL: NCT06545942
Title: A Phase 1 Study of MOMA-313 Given as Monotherapy or in Combination With a PARP Inhibitor in Participants With Advanced or Metastatic Solid Tumors
Brief Title: Study of Orally Administered MOMA-313 in Participants With Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: MOMA Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MOMA-313-001
Record Dates: First submitted 2024-07-26; First posted 2024-08-09 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumor; Metastatic Solid Tumor; Prostate Cancer; Pancreas Cancer; Breast Cancer; Ovarian Cancer; Homologous Recombination Deficiency
Keywords: Phase 1; MOMA-313; Polymerase theta; MOMA Therapeutics; Advanced Solid Tumor; Metastatic Solid Tumor; Prostate Cancer; Pancreas Cancer; Breast Cancer; Ovarian Cancer; Homologous Recombination Deficiency; HRD Mutation; Advanced (including locally)
MeSH Terms: conditions — Neoplasm Metastasis; Prostatic Neoplasms; Pancreatic Neoplasms; Breast Neoplasms; Ovarian Neoplasms | interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MOMA-313 Monotherapy (Treatment Arm 1) (Experimental): MOMA-313 administered as a single-agent in 21-day cycles.
  Interventions: Drug: MOMA-313
- MOMA-313 in Combination with Olaparib (Treatment Arm 2) (Experimental): MOMA-313 administered together with twice daily (BID) olaparib in 28-day cycles.
  Interventions: Drug: MOMA-313; Drug: Olaparib

INTERVENTIONS:
Drug: MOMA-313 — MOMA-313 administered orally
Drug: Olaparib — Olaparib administered orally
  Arms: MOMA-313 in Combination with Olaparib (Treatment Arm 2)

SUMMARY:
This Phase 1, multi-center, open-label, dose escalation and dose optimization study is designed to assess the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PDx), and preliminary clinical activity of MOMA-313 administered orally as a single agent or combination therapy in patients with homologous recombinant deficient solid tumors.

DETAILED DESCRIPTION:
MOMA-313 is a novel therapeutic agent designed to target homologous recombination (HR)-deficient cancers by inhibiting DNA polymerase theta. MOMA-313 is being developed as a single-agent and in combination with a poly (adenosine diphosphate ribose) polymerase (PARP) inhibitor in patients with HR-deficient advanced (including locally), relapsed or metastatic solid tumors.

This phase 1, first-in-human, open-label study of MOMA-313 is primarily intended to evaluate the safety and tolerability of MOMA-313 when administered orally as a single agent (Treatment Arm 1) or in combination with olaparib (Treatment Arm 2). Each treatment arm of the study includes a dose-escalation phase followed by a dose-optimization phase. In the dose-escalation phase of each treatment arm, successive cohorts of patients will receive increasing oral doses of MOMA-313 as a single agent or in combination with olaparib to determine the presumptive optimal biologic dose(s) (OBD) in this population. The dose-optimization phase of each arm will enroll additional patients to support the confirmation of the OBD.

The data from this study conducted in patients with HR-deficient advanced (including locally), relapsed or metastatic solid tumors, including safety, tolerability, PK/PDx findings, and antitumor activity, will form the basis for subsequent clinical development of MOMA-313 as a single-agent and in combination with olaparib.

ELIGIBILITY:
Key Inclusion Criteria:

1. Age ≥ 18 years
2. Have histologically confirmed disease for each treatment arm as follows:

   1. Treatment Arm 1 (MOMA-313 Monotherapy)

      - Advanced (including locally), relapsed or metastatic solid tumors that are not eligible for curative therapy, with any HR-deficient alteration.
   2. Treatment Arm 2 (MOMA-313 in Combination with Olaparib):

      * Dose escalation: Advanced (including locally), relapsed or metastatic solid tumors that are not eligible for curative therapy, for which a PARP inhibitor is indicated, with select HR-deficient mutations. Patients may be PARP inhibitor naive or exposed.
      * Dose optimization: Advanced (including locally), relapsed or metastatic CRPC or pancreatic ductal adenocarcinoma (PDAC) with select HR-deficient mutations. Patients must be PARP inhibitor naive.
3. Have at least 1 lesion at baseline (measurable or non-measurable) suitable for repeat imaging evaluation by RECIST and/or PCWG-3
4. ECOG PS ≤ 2
5. Fully recovered from clinically relevant effects of prior therapy, radiotherapy, and/or surgery **hormonal therapy allowed. Palliative radiotherapy allowed.
6. Adequate organ function per local labs
7. Comply with contraception requirements
8. Written informed consent must be obtained according to local guidelines

Key Exclusion Criteria:

1. Active prior or concurrent malignancy (some exceptions allowed)
2. Clinically relevant cardiovascular disease
3. Known CNS metastasis associated with progressive neurological symptoms (stable doses of corticosteroids allowed)
4. Known active infection
5. Prior polymerase theta inhibitor exposure
6. Known allergy, hypersensitivity, and/or intolerance to MOMA-313
7. Olaparib exposed patients with known hypersensitivity to PARP inhibitors (for patients considered for olaparib only)
8. Impaired GI function that may impact absorption.
9. Patient is pregnant or breastfeeding.
10. Known to be HIV positive, unless all of the following criteria are met:

    1. Undetectable viral load or CD4+ count ≥300 cells/μL
    2. Receiving highly active antiretroviral therapy
    3. No AIDS-related illness within the past 12 months
11. Active liver disease (some exceptions are allowed)
12. Prior or ongoing condition, therapy, or laboratory abnormality that, in the investigator's opinion, may affect safety of the patient, confound the results of the study, and/or interfere with the patients participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with AEs, dose-limiting toxicities (DLTs), serious AEs (SAEs), and/or AEs leading to discontinuation | From screening until treatment discontinuation (up to 35 months)
  To assess the safety and tolerability of MOMA-313 given as a single-agent or in combination with olaparib

SECONDARY OUTCOMES:
Identify the recommended phase 2 dose (RP2D) | From screening until treatment discontinuation (up to 35 months)
  Determine the RP2D of MOMA-313 as a single-agent or in combination with olaparib
PK parameter: area under curve (AUC) of MOMA-313 | Up to 6 weeks with sparse sampling up to 35 months
PK parameter: maximum concentration (Cmax) of MOMA-313 | Up to 6 weeks with sparse sampling up to 35 months
PK parameter: time to maximum concentration of MOMA-313 | Up to 6 weeks with sparse sampling up to 35 months
PK parameter: half-life of MOMA-313 | Up to 6 weeks with sparse sampling up to 35 months
Plasma concentration of olaparib | Up to 6 weeks with sparse sampling up to 35 months
Objective response rate (ORR) | Up to 35 months
  ORR is defined as the percentage of subjects with evidence of a complete response (CR) or partial response (PR) as per Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1 and/or Prostate Cancer Working Group-3 (PCWG-3).
Duration of response (DOR) | Up to 35 months
  DOR is defined as time from first documented PR or better to disease progression (as assessed by RECIST v1.1 and/or PCWG-3 by Investigator assessment) or death whichever is earlier for participants who have achieved a CR or PR
Time to response (TTR) | Up to 35 months
  TTR is defined as the period of time from the date of first dose of study treatment until the first objective documentation of a CR or PR per RECIST 1.1 and/or PCWG-3.
Progression free survival (PFS) | Up to 35 months
  PFS is time from first dose of study treatment to progressive disease or death from any cause, whichever is earlier, as assessed via RECIST v1.1 and/or PCWG-3 by Investigator assessment
Disease control rate (DCR) | Up to 35 months
  DCR defined by the proportion of subjects who achieved either a complete response (CR), partial response (PR), or stable disease (SD) at their first scheduled disease assessment according to disease-specific response criteria.
Overall survival (OS) | Up to 35 months
  OS is defined as the time from first dose of study treatment to the date of death, irrespective of the cause of death

CONTACTS AND LOCATIONS:
Locations (18):
- United States (12):
  - Investigative Site #108, Goodyear, Arizona
  - Investigative Site #101, La Jolla, California
  - Investigative Site #111, San Francisco, California
  - Investigative Site #104, Lake Mary, Florida
  - Investigative Site #110, St Louis, Missouri
  - Investigative Site #103, New York, New York
  - Investigative Site #106, New York, New York
  - Investigative Site #109, Philadelphia, Pennsylvania
  - Investigative Site #107, Myrtle Beach, South Carolina
  - Investigative Site #102, Nashville, Tennessee
  - Investigative Site #105, San Antonio, Texas
  - Investigative Site #112, Fairfax, Virginia
- Spain (3):
  - Investigative Site #114, Barcelona
  - Investigative Site #116, Barcelona
  - Investigative Site #115, Madrid
- United Kingdom (3):
  - Investigative Site #113, London
  - Investigative Site #117, Manchester
  - Investigative Site #118, Newcastle upon Tyne